CLINICAL TRIAL: NCT00666133
Title: Treatment Approaches for Preeclampsia in Low-Resource Settings
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Gynuity Health Projects (Other)
Collaborators: Christian Medical College, Vellore, India (Other); Chhatrapati Shahuji Maharaj Medical University (Other); Government Medical College, Nagpur (Industry); MacArthur Foundation (Other)
Responsible Party: Dr. Beverly Winikoff, President, Gynuity Health Projects
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 4.2.1
Record Dates: First submitted 2008-04-22; First posted 2008-04-24 (Estimated); Last update posted 2009-12-09 (Estimated); Status verified 2009-12

CONDITIONS: Preeclampsia
Keywords: Preeclampsia; Eclampsia; Magnesium Sulfate
MeSH Terms: conditions — Pre-Eclampsia; Eclampsia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 2 (No Intervention): Women in Group II (standard of care) will receive an 8 mL loading dose containing 4g magnesium sulfate administered manually per standard hospital protocol. The solution will be diluted with normal saline according to standard hospital practice, and given IV over 20 minutes. For women in Group II, the IV loading dose will be followed immediately with 20 mL treatment by IM injection, given as 10 mL (5 g magnesium sulfate) into each buttock. This dose will be followed by 10 mL treatments (5g magnesium sulfate) every four hours, injected into alternate buttock. Treatment will be discontinued when clinically indicated.
- 1 (Experimental): Women in Group I (Springfusor® arm) will receive a 8 mL loading dose containing 4g magnesium sulfate heptahydrate (MgSO4*7H2O) 50% solution, which is approximately 2 mmoL magnesium/mL. The loading dose of 8mL with 4 g MgSO4will be administered using the Springfusor® pump. For women in Group I, the administration of the loading dose will be immediately followed by a maintenance infusion. The maintenance dose of 4 g (8 cc, 50% MgSO4) will be administered with the Springfusor® pump continuously over four hours. The pump will be started immediately after the initial bolus and the 4g dose repeated (and syringe replaced) every four hours for upto 24 hours postpartum.
  Interventions: Device: SpringFusor Pump

INTERVENTIONS:
Device: SpringFusor Pump — Women in Group I (Springfusor® arm) will receive loading and maintenance doses of magnesium sulfate administered via an IV infusion administered with the Springfusor pump, a simple, inexpensive flow-controlled pump system.
  Arms: 1

SUMMARY:
Preeclampsia is a condition unique to pregnancy characterized by the new onset of hypertension and proteinuria. Eclampsia, characterized by maternal seizures, is a serious complication increasing the risk of maternal and infant mortality and morbidity. Magnesium sulfate is the drug of choice for prevention and treating convulsions in severe preeclampsia and eclampsia.

Magnesium sulfate is administered parenterally by intramuscular (IM) or intravenous routes (IV). In general a loading dose of 4 to 5 grams of magnesium sulfate is administered intravenously followed by an IM injection every 4 hours or by a continuous IV infusion. The IV regimen achieves more stable serum levels of magnesium but requires the use of an infusion pump for safe delivery and has a greater potential for inadvertent overdose. Although magnesium sulfate has been demonstrated as a safe and effective drug for the treatment and prevention of severe preeclampsia and eclampsia, concerns about the safety of the drug remain. The IM dosing regimen, while potentially safer, requires repeated painful IM injections. These limitations in administration hinder the widespread use of magnesium sulfate despite its demonstrated benefits.

The goal of this research is to develop a system of care that avoids overdose and facilitates the use of magnesium sulfate for the treatment of preeclampsia. To this end, a primary objective of this research is to demonstrate the safety of a simple, inexpensive flow controlled pump system (Springfusor®). This randomized study will compare the administration of magnesium sulfate by the Springfusor® controlled pump with an IM regimen, the standard of care in most hospitals in India. The study will document the efficacy and acceptability of each treatment for patients and staff and compare the cost and time elements involved in providing each method.

ELIGIBILITY:
Inclusion Criteria:

* Exhibit systolic blood pressure > 140mm Hg OR a diastolic pressure > 100 mm Hg;
* Exhibit proteinuria > 1+;
* Have not given birth, or be 24h or less postpartum;
* Exhibit urine output >100 ml or more during the previous 4h or greater than 25 mL/h;
* Agree to comply with study procedures;
* Be > 18 years of age;
* Give informed consent for study participation

Exclusion Criteria:

* Eclamptic or seizing at the time of enrollment
* Received magnesium sulfate therapy 24h prior to study enrollment

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 304 (Estimated)
Dates: Start 2008-04; Primary Completion 2009-10 (Actual); Study Completion 2009-10 (Actual)

PRIMARY OUTCOMES:
completed course of treatment | 24 hours postpartum

CONTACTS AND LOCATIONS:
Overall Officials: Beverly Winikoff, MD, MPH, Principal Investigator — Gynuity Health Projeccts
Locations (2):
- India (2):
  - Government Medical College, Nagpur, Maharashtra
  - Christian Medical College, Vellore, Tamil Nadu

REFERENCES:
- [Derived] Salinger DH, Mundle S, Regi A, Bracken H, Winikoff B, Vicini P, Easterling T. Magnesium sulphate for prevention of eclampsia: are intramuscular and intravenous regimens equivalent? A population pharmacokinetic study. BJOG. 2013 Jun;120(7):894-900. doi: 10.1111/1471-0528.12222. Epub 2013 Mar 26. PMID 23530757